CLINICAL TRIAL: NCT07402538
Title: SBRT Followed by Neoadjuvant Chemoimmunotherapy Before Surgery in Resectable Locally Advanced Oral and HPV-unrelated Oropharyngeal Squamous Cell Carcinoma: a Randomized Controlled Phase III Trial
Brief Title: Surgery With or Without Neoadjuvant Treatment of SBRT Plus Chemoimmunotherapy in Resectable Locally Advanced Oral and HPV-unrelated Oropharyngeal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-532-X01
Record Dates: First submitted 2026-01-16; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Oral Cancer; Oropharyngeal Cancer
Keywords: SBRT; neoadjuvant therapy; locally advanced oral/oropharyngeal cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — Chemoradiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant treatment followed by surgery arm (Experimental): Initially, the patient underwent neoadjuvant treatment, including stereotactic body radiotherapy (SBRT) followed by chemoimmunotherapy of Tislelizumab (200 mg), Docetaxel (75 mg/m²), and Cisplatin (75 mg/m²). A subsequent imaging re-examination is to be performed for assessment two weeks after the last chemotherapy cycle. Finally, curative surgical resection should be performed 3-4 weeks after the last chemotherapy cycle, followed by adjuvant postoperative radiotherapy or chemoradiotherapy.
  Interventions: Combination Product: Neoadjuvant treatment of SBRT plus chemoimmunotherapy followed by surgery and postoperative radiotherapy or chemoradiotherapy
- Surgery arm (Active Comparator): Radical surgery followed by postoperative radiotherapy or chemoradiotherapy.
  Interventions: Combination Product: Surgery and postoperative radiotherapy or chemoradiotherapy

INTERVENTIONS:
Combination Product: Neoadjuvant treatment of SBRT plus chemoimmunotherapy followed by surgery and postoperative radiotherapy or chemoradiotherapy — The patient was initially subjected to a neoadjuvant treatment regime, encompassing stereotactic body radiotherapy (SBRT) and chemoimmunotherapy. The SBRT was administered with a dose of 6 Gy per fraction to the primary tumour and metastatic lymph nodes, administered every other day for a total of three fractions. Following this, a period of one to two weeks was to elapse before the initiation of Tislelizumab (200 mg), Docetaxel (75 mg/m²), and Cisplatin (75 mg/m²), on a three-week cycle, for a total of two cycles. A subsequent imaging re-examination was to be performed for assessment two weeks after the final chemotherapy cycle. Finally, curative surgical resection was to be performed 3-4 weeks after the final chemotherapy cycle, followed by adjuvant postoperative radiotherapy or chemoradiotherapy with cisplatin at a dose of 100 mg/m² for two cycles.
  Arms: Neoadjuvant treatment followed by surgery arm
Combination Product: Surgery and postoperative radiotherapy or chemoradiotherapy — Radical surgery followed by postoperative radiotherapy or chemoradiotherapy with cisplatin at a dose of 100 mg/m² for three cycles.
  Arms: Surgery arm

SUMMARY:
The objective of this study is to evaluate the efficacy of neoadjuvant stereotactic body radiation therapy (SBRT) in combination with chemotherapy and immunotherapy, prior to radical surgery, in enhancing the 2-year event-free survival rate and overall survival rate in patients diagnosed with locally advanced oral or HPV-unrelated oropharyngeal cancer.

ELIGIBILITY:
The inclusion criteria for this study are as follows:

* Histologically and/or cytologically confirmed treatment-naïve oral squamous cell carcinoma or HPV-negative oropharyngeal squamous cell carcinoma.
* Clinical stage III -Ⅳa (8th edition of AJCC).
* Age: 18 to 75 years old.
* According to the Eastern Cooperative Oncology Group (ECOG) criteria (with a performance status score of 0 or 1).
* Good organ function.
* Expected survival time: ≥ 3 months.
* The patient has signed the informed consent form and is willing and able to comply with the study's scheduled visits, treatment plans, laboratory tests, and other research procedures.
* Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrolment and must agree to use highly effective contraceptive measures during the study period and for at least 60 days after the last dose (including chemotherapeutic drugs and Tislelizumab).
* If the female partner of a male subject is still of childbearing potential, the male subject must agree to use highly effective contraceptive measures during the study period and for at least 60 days after the last dose.

Exclusion Criteria:

* Patients with concurrent other malignant tumors
* Patients with known or suspected autoimmune diseases, including dementia and epilepsy.
* Patients with severe mental disorders at the same time
* Patients with necrotic lesions who are assessed by the investigator as having a risk of massive hemorrhage
* Patients with severe heart disease or pulmonary dysfunction, and those with cardiac or pulmonary function grade ≤ 3 (grade 3 inclusive)
* Patients with laboratory test results that do not meet the relevant criteria within 7 days prior to enrollment
* Received systemic or local glucocorticoid therapy within 4 weeks prior to enrollment
* Patients with comorbidities requiring long-term treatment with immunosuppressive drugs, or requiring systemic or local administration of corticosteroids at immunosuppressive doses.
* Patients with active tuberculosis (TB), who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year prior to screening.
* A history of prior use of anti-Tislelizumab, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-CTLA-4 antibodies (or any other antibodies targeting T-cell co-stimulation or checkpoint pathways).
* Subjects with any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism); subjects with vitiligo or those whose childhood asthma has been completely relieved and who do not require any intervention in adulthood are eligible for enrollment; those with asthma requiring medical intervention with bronchodilators are not eligible for enrollment.
* HIV-positive subjects
* Positive for HBsAg with concurrent positive HBV DNA copy number (quantitative test ≥ 1000 cps/ml); positive for chronic hepatitis C on blood screening (HCV antibody positive)
* Received any anti-infective vaccines (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment
* Pregnant women with positive pregnancy test results among females of childbearing potential and lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to two years.
  The time interval from randomization to the occurrence of imaging tumor progression during the neoadjuvant treatment stage that makes surgery impossible, or postoperative imaging or biopsy results show local tumor recurrence, lymph node recurrence, distant metastasis, or death for any cause.

SECONDARY OUTCOMES:
2-year overall survival | From date of randomization until the date of death from any cause, assessed up to two years.
  The time interval from random start to death for any cause.
MPR | Three weeks after surgery
  Proportion of patients with ≤10% viable tumor cells identified per AJCC/CAP Tumor Regression Grading (TRG) protocol evaluation of surgical specimens.
pCR | Three weeks after surgery
  Proportion of patients with no viable tumor cells identified upon complete and systematic evaluation of postoperative specimens under the AJCC/CAP Tumor Regression Grading (TRG) protocol, including microscopic examination of all sampled primary tumor sites and regional lymph nodes.
Mandibular Preservation Rate | On the day of surgery
  Proportion of oral cancer patients retaining mandibular continuity after primary tumor resection.
Incidence rates of AEs (Adverse Events) and SAEs (Serious Adverse Events) | Through study completion, an average of 3 year
  Percentage of patients with adverse events ≥ Grade 3 among all treated patients.
Quality of life assessment | Postoperatively at 24 months
  Quality of life was assessed using the EORTC QLQ-C30 scale at postoperative time point of 2 year.
Quality of life assessment | Postoperatively at 24 months
  Quality of life was assessed using the QLQ-H&N35 scale at postoperative time point of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Yun Xie, M.D., Principal Investigator — Sun Yat-sen University; Ming Song, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No